CLINICAL TRIAL: NCT05252936
Title: Effectiveness of a Mayan Language Social Media Campaign on COVID-19 Vaccine
Brief Title: Effectiveness of a Mayan Language Social Media Campaign on COVID-19 Vaccine Beliefs in Guatemala
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Wuqu' Kawoq, Maya Health Alliance (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Jamie Johnston, Research Director, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 63193
Record Dates: First submitted 2022-02-21; First posted 2022-02-23 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Vaccination Refusal
MeSH Terms: conditions — Vaccination Refusal

STUDY DESIGN:
Intervention Model Description: To investigate the effectiveness of Mayan language content, we are testing three treatment arms - visually identical videos in the 1) Spanish language, 2) K'iche' language, and 3) Kaqchikel language. We will measure effects of the three treatment arms across Spanish speakers (including K'iche' and Kaqchikel speakers who also speak Spanish). We will also measure the effectiveness of K'iche vs. Spanish content among K'iche speakers and Kaqchikel vs. Spanish content for Kaqchikel speakers.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Spanish language content (Experimental): Social media campaign content with Spanish language voiceover
  Interventions: Other: COVID-19 vaccine social media campaign exposure
- K'iche' language content (Experimental): Social media campaign content with K'iche' language voiceover
  Interventions: Other: COVID-19 vaccine social media campaign exposure
- Kaqchikel language content (Experimental): Social media campaign content with Kaqchikel language voiceover
  Interventions: Other: COVID-19 vaccine social media campaign exposure
- Control (Active Comparator): A control group that is not exposed to any of the social media campaign content will serve as control to allow for comparison of outcomes with treatment arms.
  Interventions: Other: COVID-19 vaccine social media campaign exposure

INTERVENTIONS:
Other: COVID-19 vaccine social media campaign exposure — A series of animated video clips will be promoted through Facebook Ads and randomized at the individual level across Facebook users throughout the entire country. To investigate the effectiveness of Mayan language content, we are testing three treatment arms - visually identical videos in the 1) Spanish, 2) K'iche', and 3) Kaqchikel languages. The videos are visually identical and follow the same audio script, translated into the three focal language. Local voiceover artists were used to record the scripts in the three languages. A control group that is not exposed to any of the social media campaign content will serve as active comparator to allow for comparison of outcomes with treatment arms.

SUMMARY:
Prior evidence, including formative work supporting the development of this study, suggests there is widespread vaccine hesitancy among Indigenous communities in Guatemala, fueled by mistrust in the health system, lack of official information, and the circulation of myths and misinformation. We will test the effectiveness of a video-based social media campaign that provides a basic overview of the science behind COVID-19 vaccines and addresses prevalent myths and misinformation being shared in target communities. A series of animated videos will be promoted through Facebook Ads and randomized at the individual level across Facebook users throughout the entire country. To investigate the effectiveness of Mayan language content, we are testing three treatment arms - visually identical videos in the 1) Spanish language, 2) K'iche' language, and 3) Kaqchikel language. Our primary outcomes are responses to two attitudinal questions collected via Facebook polling: 1) How safe do you think a COVID-19 vaccine is for people like you? (options: very safe, somewhat safe, barely safe, not safe, don't know); and 2) When you think of most people whose opinion you value, how much would they approve of people getting a COVID-19 vaccine? (options: definitely approve, mostly approve, somewhat approve, not at all approve, don't know). We will measure effects of the three treatment arms across Spanish speakers (including K'iche' and Kaqchikel speakers who also speak Spanish). We will also measure the effectiveness of K'iche vs. Spanish content among K'iche speakers and Kaqchikel vs. Spanish content for Kaqchikel speakers.

ELIGIBILITY:
Inclusion Criteria:

* The intervention will be delivered through the Facebook Ads platform. Intervention content will be promoted to Facebook Users throughout the entire country of Guatemala. K'iche' content will be targeted only in departments where the K'iche' language is primarily spoken. Kaqchikel content will be targeted only in departments where the Kaqchikel language is primarily spoken.

Exclusion Criteria:

* Only adult Facebook users of age 18 will be included. Users under age 18 are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 5000 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Beliefs about COVID-19 vaccine safety | 4 weeks
  Our primary outcomes are responses to two attitudinal questions collected via Facebook polling. This outcome is response to the question: How safe do you think a COVID-19 vaccine is for people like you? (options: very safe, somewhat safe, barely safe, not safe, don't know).
Beliefs about COVID-19 vaccine acceptance among social network | 4 weeks
  Our primary outcomes are responses to two attitudinal questions collected via Facebook polling. This outcome is response to the question: When you think of most people whose opinion you value, how much would they approve of people getting a COVID-19 vaccine? (options: definitely approve, mostly approve, somewhat approve, not at all approve, don't know).

CONTACTS AND LOCATIONS:
Locations (1):
- Wuqu' Kawoq - Maya Health Alliance, Tecpán Guatemala, Guatemala

IPD SHARING:
Plan to Share IPD: No